CLINICAL TRIAL: NCT03170375
Title: Dietary Prevention of Heart Failure in Hypertensive Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: CARA-009-16F; 9050 (Other Grant/Funding Number: VA CSR&D Merit)
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
Keywords: obesity; sodium; DASH diet; hypertension; vascular stiffness; diastolic function
MeSH Terms: conditions — Heart Failure; Obesity; Hypertension | interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: Phase 1 of study: sequential design, 14 days each of usual diet followed by 14 days of sodium-restricted DASH diet Phase 2 of study: randomized assignment, 6 months of motivational interviewing vs. motivational interviewing plus mobile application-based promotion of dietary adherence
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational Interviewing + WHEELS-I (Experimental): In addition to motivational interviewing-based counseling with a registered dietitian to promote adoption of the sodium-restricted Dietary Approaches to Stop Hypertension (DASH/SRD) eating plan., participants in this arm will also receive an electronically-delivered tailored messaging intervention called Women's and Men's Hypertension Experiences and Emerging Lifestyle Intervention (WHEELS-I). Randomization will occur after phase 1 of the study which includes 2 weeks of an ad lib diet followed by 2 weeks of prepared pre-packaged DASH/SRD meals.
  Interventions: Behavioral: Performance of WHEELS-I in promoting DASH/SRD adoption
- Motivational Interviewing (Active Comparator): Participants in this arm will receive motivational interviewing-based counseling with a registered dietitian to promote adoption of the sodium-restricted Dietary Approaches to Stop Hypertension (DASH/SRD) eating plan. Randomization will occur after phase 1 of the study which includes 2 weeks of an ad lib diet followed by 2 weeks of prepared pre-packaged DASH/SRD meals.
  Interventions: Behavioral: Performance of WHEELS-I in promoting DASH/SRD adoption

INTERVENTIONS:
Behavioral: Performance of WHEELS-I in promoting DASH/SRD adoption — All participants will receive motivational interviewing (MI) based counseling. Participants in the MI + WHEELS-I arm will also receive the WHEELS-I electronically-delivered tailored messaging.
  Other Names: Phase 2

SUMMARY:
Tens of thousands of Veterans have heart failure with preserved ejection fraction (HFpEF), and suffer poor quality of life, frequent hospitalizations, and high death rates. Older Veterans and those with high blood pressure, obesity, and the metabolic syndrome (abnormal cholesterol and resistance to insulin's effects) are particularly at risk for HFpEF. However, it is not clear why only some Veterans in this risk group eventually develop HFpEF. Extensive information from experimental animal models and some human studies suggests that dietary patterns in vulnerable 'salt-sensitive' people could contribute to the risk for HFpEF. Reducing salt intake and increasing overall dietary quality in at-risk Veterans could prevent heart and blood vessel damage that ultimately leads to HFpEF. Reducing the development of HFpEF, which currently has no definitive treatment, is highly relevant to the VA's mission to emphasize prevention of disease and population health.

DETAILED DESCRIPTION:
COVID-19 in-person visit hold has been removed- screening and actively enrolling. We are not currently performing sublingual darkfield microscopy because of the need for close face-to-face contact with an open-mouthed patient for several minutes in the setting of COVID-19 pandemic.

Patients with heart failure (HF) account for over 1,200,000 VA outpatient visits per year, and HF remains the most common cause for hospital admission in the VA. Approximately 1/3 of Veterans with HF have 'preserved' ejection fraction (HFpEF), or relatively normal contractile function of the heart; such patients suffer functional decline and poor quality of life, and half die within 5 years after diagnosis. Risk factors for developing HFpEF are more common in Veterans than the general population, and the burden of HFpEF to the VA system will rise in the years ahead as these Veterans age. Preventive efforts are critical, but are hampered by gaps in knowledge related to HFpEF pathophysiology. The long term goal of this proposal is to prevent the onset of HFpEF in at-risk Veterans. Hypertension (HTN) confers the highest population-attributable risk for HFpEF, particularly when accompanied by the metabolic syndrome, a constellation of obesity, insulin resistance, and dyslipidemia. Animal models of HTN and metabolic syndrome develop HFpEF due to microvascular oxidative stress and inflammation induced by high sodium intake. Recent data from cardiac biopsies confirm similar mechanisms in human HFpEF. Dietary sodium restriction is widely recommended to prevent HTN-associated heart disease in humans, but this advice is now controversial. Few studies have examined how individual differences in response to sodium intake affect risk. "Salt-sensitive" persons have blood pressure (BP) that changes in parallel with sodium intake, and commonly develop cardiovascular abnormalities associated with HFpEF. The overall objective of this proposal is to evaluate salt-sensitivity as a novel, diet-responsive risk factor for incident HFpEF in Veterans with HTN and metabolic syndrome. The central hypothesis is that the sodium-restricted Dietary Approaches to Stop Hypertension (DASH/SRD) eating pattern will improve cardiovascular functional and structural risk factors for HFpEF in Veterans with the salt-sensitive phenotype. Guided by findings in experimental models, cohort studies, and strong preliminary evidence from the investigators' research group, this hypothesis will be tested in a two-phase study and by pursuing three specific aims: 1) Determine effects of DASH/SRD on functional and structural cardiovascular HFpEF risk factors in salt-sensitive vs. salt-resistant Veterans, 2) measure the effect of an electronically-delivered tailored-messaging intervention on DASH/SRD adherence, and 3) determine effects of DASH/SRD intervention and adoption on microvascular function and assess the endothelial glycocalyx as a biomarker of cardiovascular response to DASH/SRD. Phase 1 of the study is a sequential comparison of DASH/SRD vs. control diet for two weeks each, and Phase 2 a 6-month extension to promote DASH/SRD adherence. The salt-sensitive phenotype will be defined by between-diet changes in 24-hour mean BP during Phase 1. In Phase 2, the efficacy of motivational interviewing-based counseling and the Women's and Men's Hypertension Experiences and Emerging Lifestyles Intervention (WHEELS-I), a tailored messaging program, to sustain DASH/SRD adherence, will be compared. Echocardiography and arterial tonometry will be used to assess HFpEF-related cardiovascular parameters during short- and longer-term dietary modification and their interaction with salt-sensitivity. In vivo microscopy and novel blood testing will assess microvascular function and the integrity of the endothelial glycocalyx, a blood vessel lining that is sodium-responsive and may mediate the adverse effects of salt-sensitivity. This proposal is innovative because it represents the first study to examine salt-sensitivity as a factor promoting HFpEF in Veterans with HTN and metabolic syndrome, the highest risk group for incident HFpEF. Moreover, it aims to link microvascular dysfunction, an important pathway in human HFpEF, with endothelial glycocalyx damage, a potential biomarker for sodium-mediated vascular risk. The proposed research is significant because it will vertically advance the investigators' understanding of how dietary factors contribute to the pathophysiology of HFpEF, a major and growing health threat to Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 45 years with HTN

  * here defined as screening systolic BP 130 and/or diastolic BP 85 mmHg, or current use of anti-hypertensive drugs
* and metabolic syndrome

  * body mass index 30 kg/m2 and/or waist circumference >94 cm
* Participants must also be willing to participate in the WHEELS-I program by using a smartphone application or email

Exclusion Criteria:

* On-treatment systolic BP of >160 mmHg at screening visit
* previous history of HF
* left ventricular ejection fraction <50%
* moderate or severe valvular heart disease
* myocardial infarction or stroke within the prior 6 months
* chronic kidney disease with estimated glomerular filtration rate <45 ml/min/ 1.73m2
* unoperated aortic aneurysm for which surgery is indicated, prior hyperkalemia requiring urgent treatment
* hemoglobin <9 gm/dL
* investigator-determined factors: severe pulmonary disease, e.g.:

  * oxygen-requiring
* hepatic disease, e.g.:

  * cirrhosis
* severely uncontrolled diabetes (hemoglobin A1c >10%)
* active cancer other than non-melanoma skin or low-risk prostate cancer
* other comorbidity with expected survival <12 months
* active alcohol/illicit substance abuse
* and/or a history of persistent nonadherence to treatment
* Veterans involved in another study (unless it is survey-only and the other investigator will allow us to invite the person in a survey-only study to consider our study)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott L. Hummel, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1:
  Screening visit: Follow baseline diet for 2 weeks Excluded if patient couldn't wean from renin-angiotensin-aldosterone system (RAAS) inhibitors and diuretics without complications
  2-week visit: follow DASH-SRD diet for 2 weeks
  4-week visit: randomized into Arm 1 or 2 and begin phase II of study.
Groups:
- Phase 1: 2-week Diet As Usual Then 2 Weeks of DASH/SRD Diet: Consented participants will have clinic BP measured at the screening visit and will enter a two-week usual diet period, during which antihypertensive medications, with the exception of calcium channel blockers, will be weaned off. During this time period, the participant will consume their usual diet. Following the usual diet period and the week 2 visit, participants will consume the DASH/SRD diet for 14 days each.
- Motivational Interviewing + WHEELS-I: In addition to motivational interviewing-based counseling with a registered dietitian to promote adoption of the sodium-restricted Dietary Approaches to Stop Hypertension (DASH/SRD) eating plan., participants in this arm will also receive an electronically-delivered tailored messaging intervention called Women's and Men's Hypertension Experiences and Emerging Lifestyle Intervention (WHEELS-I). Randomization will occur after phase 1 of the study which includes 2 weeks of an ad lib diet followed by 2 weeks of prepared pre-packaged DASH/SRD meals.
  Performance of WHEELS-I in promoting DASH/SRD adoption: Participants will receive the WHEELS-I electronically-delivered tailored messaging intervention in addition to motivational interviewing-based counseling.
Period: Phase 1 - 4 Weeks
Arm/Group | Phase 1: 2-week Diet As Usual Then 2 Weeks of DASH/SRD Diet | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Started | 71 | 0 | 0
Completed | 66 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0
Period: Phase 2 - 6 Months
Arm/Group | Phase 1: 2-week Diet As Usual Then 2 Weeks of DASH/SRD Diet | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Started | 0 | 28 | 38
Completed | 0 | 25 | 36
Not Completed | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: The population for baseline analysis includes all 71 participants who started in Phase 1, which includes the 66 participants who continued into the randomization phase.
Groups:
- Phase 1: 2-week Diet As Usual Then 2 Weeks of DASH/SRD Diet: This arm includes all participants who started Phase 1 of the study. Phase 1 took place prior to randomization into either the Motivational Interviewing or Motivational Interviewing + WHEELS-I arm.
- Total: Total of all reporting groups
Arm/Group | Phase 1: 2-week Diet As Usual Then 2 Weeks of DASH/SRD Diet | Motivational Interviewing + WHEELS-I | Motivational Interviewing | Total
Number analyzed (Participants) | 71 | 28 | 38 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  years
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1 | 66 (8) |  |  | 66 (8)
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2 |  | 64 (9) | 67 (8) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants] — Data collected from Phase 1 and Phase 2 are reported in separate Rows Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  Participants
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1: Female | 11 |  |  | 11
    Phase 1: Male | 60 |  |  | 60
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2: Female |  | 3 | 7 | 10
    Phase 2: Male |  | 25 | 31 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  Participants
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1: Hispanic or Latino | 4 |  |  | 4
    Phase 1: Not Hispanic or Latino | 63 |  |  | 63
    Phase 1: Unknown or Not Reported | 4 |  |  | 4
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2: Hispanic or Latino |  | 3 | 0 | 3
    Phase 2: Not Hispanic or Latino |  | 23 | 36 | 59
    Phase 2: Unknown or Not Reported |  | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  Participants
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1: American Indian or Alaska Native | 0 |  |  | 0
    Phase 1: Asian | 1 |  |  | 1
    Phase 1: Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
    Phase 1: Black or African American | 10 |  |  | 10
    Phase 1: White | 57 |  |  | 57
    Phase 1: More than one race | 0 |  |  | 0
    Phase 1: Unknown or Not Reported | 3 |  |  | 3
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2: American Indian or Alaska Native |  | 0 | 0 | 0
    Phase 2: Asian |  | 1 | 0 | 1
    Phase 2: Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0
    Phase 2: Black or African American |  | 2 | 8 | 10
    Phase 2: White |  | 23 | 29 | 52
    Phase 2: More than one race |  | 0 | 0 | 0
    Phase 2: Unknown or Not Reported |  | 2 | 1 | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  kg/m^2
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1 | 34.4 (5.1) |  |  | 34.4 (5.1)
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2 |  | 34.7 (4.7) | 34.4 (5.5) | 34.5 (5.1)
Waist Circumference [Mean (Standard Deviation); unit: cm] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  cm
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1 | 116 (14) |  |  | 116 (14)
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2 |  | 117 (9) | 116 (17) | 116 (14)
Hip Circumference [Mean (Standard Deviation); unit: cm] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  cm
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1 | 117 (15) |  |  | 117 (15)
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2 |  | 118 (11) | 116 (17) | 117 (15)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  mmHg
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1 | 133 (15) |  |  | 133 (15)
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2 |  | 136 (14) | 132 (16) | 134 (15)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  mmHg
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1 | 72 (11) |  |  | 72 (11)
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2 |  | 74 (11) | 72 (11) | 73 (11)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  mg/dL
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1 | 163 (107) |  |  | 163 (107)
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2 |  | 157 (54) | 157 (131) | 157 (105)
HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  mg/dL
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1 | 45 (10) |  |  | 45 (10)
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2 |  | 43 (9) | 46 (11) | 45 (10)
Hemoglobin A1c [Mean (Standard Deviation); unit: %] — Population: Data collected from Phase 1 and Phase 2 are reported in separate Rows
  %
    Phase 1: number analyzed (Participants) | 71 | 0 | 0 | 71
    Phase 1 | 6.2 (1.1) |  |  | 6.2 (1.1)
    Phase 2: number analyzed (Participants) | 0 | 28 | 38 | 66
    Phase 2 |  | 6.3 (1.0) | 6.3 (1.1) | 6.3 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Carotid-femoral Pulse Wave Velocity
Description: Phase 1 primary hypothesis: greater reduction in carotid-femoral pulse wave velocity with DASH diet in individuals with salt-sensitive blood pressure
  Change in velocity of pulse wave traveling between carotid and femoral artery; validated measure of arterial stiffness
Time Frame: Phase 1 of study, change between week 2 and week 4
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Salt-sensitive Participants; Non Salt-sensitive Participants: Participants are defined as having a salt-sensitive blood pressure phenotype if they have >= 4 mmHg change in mean arterial pressure by 24-hour monitoring between baseline and low-sodium diet conditions
Arm/Group | Salt-sensitive Participants | Non Salt-sensitive Participants
Number analyzed (Participants) | 28 | 31
m/s | -0.3 (1.6) | 0.4 (3.0)
Statistical Analysis 1: Comparison: Salt-sensitive Participants vs Non Salt-sensitive Participants; Test type: Superiority; p = 0.28, Regression, Linear; adjusted for baseline carotid-femoral pulse wave velocity

2. Primary Outcome: Left Ventricular Mass Index
Description: Left ventricular mass indexed to body surface area.
  Larger/greater left ventricular mass index is associated with increased long-term risk of cardiovascular events, including the development of heart failure. Normal values for men are 49-115 g/m² and for women 43-95 g/m²
Time Frame: Phase 2 of study, change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: g/m2
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Number analyzed (Participants) | 25 | 35
g/m2 | -3.3 (15.5) | -1.7 (12.2)
Statistical Analysis 1: Comparison: Motivational Interviewing + WHEELS-I vs Motivational Interviewing; Test type: Superiority; p = 0.60, Regression, Linear; adjusted for baseline left ventricular mass index

3. Secondary Outcome: Global Longitudinal Left Ventricular Strain
Description: Global longitudinal left ventricular strain (GLS), a sensitive measure of ventricular systolic function
  GLS is calculated by dividing the reduction in length of a myocardial (heart) segment from the end of diastole (maximum relaxation) to the end of systole (maximum contraction) by the segment's original length at end-diastole (i.e. change in length/original length). GLS is averaged across six myocardial segments, is expressed in a percentage, and is negative by convention since cardiac segment length decreases during systole. The more negative/greater magnitude, the better the GLS.
  Normal GLS is -18% to -22%. Low GLS is associated with long-term increased risk of cardiovascular events, including the development of heart failure.
Time Frame: Phase 1 of study, change between week 2 to week 4
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Non-salt Sensitive Participants: Participants are defined as having a salt-sensitive blood pressure phenotype if they have >= 4 mmHg change in mean arterial pressure by 24-hour monitoring between baseline and low-sodium diet conditions
Arm/Group | Salt-sensitive Participants | Non-salt Sensitive Participants
Number analyzed (Participants) | 19 | 24
ratio | -0.2 (2.5) | -0.5 (2.0)
Statistical Analysis 1: Comparison: Salt-sensitive Participants vs Non-salt Sensitive Participants; Test type: Superiority; p = 0.27, Regression, Linear; adjusted for baseline global left ventricular longitudinal strain

4. Secondary Outcome: Carotid-femoral Pulse Wave Velocity
Description: Velocity of pulse wave traveling between carotid and femoral artery; validated measure of arterial stiffness
Time Frame: Phase 2 of study, change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Number analyzed (Participants) | 23 | 34
m/s | 1.1 (1.5) | 0.3 (1.9)
Statistical Analysis 1: Comparison: Motivational Interviewing + WHEELS-I vs Motivational Interviewing; Test type: Superiority; p = 0.03, Regression, Linear; adjusted for baseline carotid-femoral pulse wave velocity

5. Other Pre Specified Outcome: Salt-sensitivity Phenotype
Description: Salt-sensitive blood pressure means that blood pressure changes more than 'normal' when dietary sodium intake changes, i.e. increases or decreases in parallel with sodium intake. Having a salt-sensitive blood pressure pattern is an independent long-term risk factor for cardiovascular events. Variable testing approaches, blood pressure thresholds, and methods of blood pressure measurement have been proposed in the literature to define blood pressure salt-sensitivity.
  In this study, we report "salt-sensitive" vs. "non salt-sensitive" as a binary variable. Change in 24-hour mean blood pressure of >= 4 mmHg between the ad-lib and home-delivered meal periods of Phase 1 defines the salt-sensitive blood pressure phenotype
Time Frame: Phase 1 of study, change between week 2 and week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Number analyzed (Participants) | 25 | 38
Participants | 9 | 22

6. Other Pre Specified Outcome: 24-hour Urinary Sodium Excretion
Description: Measure of daily dietary sodium intake
Time Frame: Phase 2 of study, change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mg/24h
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Number analyzed (Participants) | 25 | 36
mg/24h | -456 (2077) | -204 (1721)

7. Other Pre Specified Outcome: Sodium-restricted DASH Diet Adherence by Food Frequency Questionnaire (FFQ)
Description: Sodium-restricted DASH diet score on FFQ, measured by quintiles of intake in 8 dietary domains as compared with age- and sex-matched norms from NHANES national US survey data. Score ranges 8-40 points, with higher scores indicating greater adherence
Time Frame: Phase 2 of study, change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Number analyzed (Participants) | 25 | 36
points | 1.5 (3.1) | 1.4 (2.8)

8. Other Pre Specified Outcome: Sodium-restricted DASH Diet Adherence
Description: Analysis of 3-day food diaries by a Registered Dietitian, utilizing the Nutrition Data System for Research. DASH diet adherence score based on proportion of recommended daily intake in 9 domains, score ranges 0-9 points with higher scores indicating greater adherence
Time Frame: Phase 2 of study, change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Number analyzed (Participants) | 23 | 35
points | 0.3 (1.3) | 0.6 (1.6)
Statistical Analysis 1: Comparison: Motivational Interviewing + WHEELS-I vs Motivational Interviewing; Test type: Superiority; p = 0.47, generalized estimating equations; Model includes time (baseline, phase 2 month 1, phase 2 month 6), randomization assignment, and time x randomization assignment

9. Other Pre Specified Outcome: Clinic Systolic Blood Pressure
Description: Change in systolic blood pressure obtained in clinic with automated brachial cuff
Time Frame: Phase 2 of study, change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Number analyzed (Participants) | 25 | 36
mmHg | -5.4 (12.9) | -4.1 (15.8)
Statistical Analysis 1: Comparison: Motivational Interviewing + WHEELS-I vs Motivational Interviewing; Test type: Superiority; p = 0.28, generalized estimating equation; [statistical method as in outcome 8, analysis 1]

10. Other Pre Specified Outcome: Clinic Diastolic Blood Pressure
Time Frame: Phase 2 of study, change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Number analyzed (Participants) | 25 | 36
mmHg | -3.2 (10.7) | -3.5 (10.8)
Statistical Analysis 1: Comparison: Motivational Interviewing + WHEELS-I vs Motivational Interviewing; Test type: Superiority; p = 0.43, generalized estimating equations; [statistical method as in outcome 8, analysis 1]

11. Other Pre Specified Outcome: Triglycerides
Description: Serum triglyceride changes during dietary intervention
Time Frame: Phase 2 of study, change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Number analyzed (Participants) | 25 | 36
mg/dL | 41 (39) | 39 (127)
Statistical Analysis 1: Comparison: Motivational Interviewing + WHEELS-I vs Motivational Interviewing; Test type: Superiority; p = 0.94, t-test, 2 sided

12. Other Pre Specified Outcome: Urine Sodium and Potassium Ratios
Description: Unitless ratio of urine sodium (in mmol) divided by urine potassium (in mmol), measured from spot samples taken from 24-hour urine samples.
Time Frame: Phase 2 of study, change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
Number analyzed (Participants) | 25 | 36
ratio | -1.2 (1.1) | -1.2 (1.2)
Statistical Analysis 1: Comparison: Motivational Interviewing + WHEELS-I vs Motivational Interviewing; Test type: Superiority; p = 0.90, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline to end of study, an average of 1 year
Groups:
- Motivational Interviewing + WHEELS-I: In addition to motivational interviewing-based counseling with a registered dietitian to promote adoption of the sodium-restricted Dietary Approaches to Stop Hypertension (DASH/SRD) eating plan, participants in this arm will also receive an electronically-delivered tailored messaging intervention called Women's and Men's Hypertension Experiences and Emerging Lifestyle Intervention (WHEELS-I). Randomization will occur after phase 1 of the study which includes 2 weeks of an ad lib diet followed by 2 weeks of prepared pre-packaged DASH/SRD meals.
Arm/Group | Motivational Interviewing + WHEELS-I | Motivational Interviewing
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/28 | 2/38
Other Adverse Events (participants affected / at risk) | 0/28 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Motivational Interviewing + WHEELS-I (N=28) | Motivational Interviewing (N=38)
Atrial fibrillation (Cardiac disorders) | 0 | 1 — Participant hospitalization and received new diagnosis of atrial fibrillation. Started on new medication and follow-up with cardiologist.
Lobectomy (Surgical and medical procedures) | 0 | 1 — Lobectomy procedure d/t lung cancer
Tooth infection (Infections and infestations) | 1 | 0 — Hospitalization for infected tooth post extraction

LIMITATIONS AND CAVEATS:
1. recruitment initially delayed 1 yr due to VA privacy/information security review for app

   Due to COVID-19:
2. no sublingual darkfield microscopy performed
3. lost 1.5 yrs recruitment time, had to decrease in-person visits

   Related to study diet:
4. Meal company changed meal offerings and no longer offered high-sodium option

Due to 3) and 4) above: changed protocol to 2 weeks ad-lib diet then 2 weeks low-sodium DASH diet Due to 1) and 3) above: unable to recruit full intended cohort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT03170375/Prot_001.pdf
  • Statistical Analysis Plan (2025-05-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT03170375/SAP_002.pdf
  • Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT03170375/ICF_000.pdf